CLINICAL TRIAL: NCT01541033
Title: Biomarker Discovery In Children With Autism Plus Familial Autoimmune History
Brief Title: Biomarker of Children With Familial Autoimmune History
Status: Completed | Type: Observational
Sponsor: Le Bonheur Children's Hospital (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Principal Investigator, James W. Wheless, Departmental Chair, Le Bonheur Children's Hospital
Other Study IDs: 08-00206-XP
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Autism; Children
Keywords: autism; children
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Autism with FAH: Children diagnosed with autism with first degree relatives that have autoimmune disorders.
- Autism without FAH: Children diagnosed with autism without first degree relatives that have autoimmune disorders.
- Control: Typically developing children

SUMMARY:
The purpose of this study is to identify biomarkers in this subset of autism patients, design a protein based assay system for screening serum for these biomarkers and confirm that these serum antibodies are still present at one year's time.

DETAILED DESCRIPTION:
Purpose: To identify biomarkers in this subset of autism patients, design a protein based assay system for screening serum for these biomarkers and confirm that these serum antibodies are still present at one year's time.

Rationale: Autistic spectrum disorders (ASD), are an increasingly important public health concern. Estimates of prevalence of ASDs range from 1/500 to 1/150 children. Retrospective data points to immune dysfunction in some of these children and increased frequency of familial autoimmune history (FAH) has been reported in children with autism. Behavioral responses to immune modulating therapy, though in uncontrolled studies, indicate a role for autoimmunity in the pathogenesis. Preliminary prospective work has suggested an immune etiology in autism based on the high frequency of brain endothelial antibodies (BEA) in children with language regression, 2/3 of whom are on the autistic spectrum and with autism without language regression. Follow up studies in a small number of patients showed persistence of BEA after at least a year. The specific nervous system epitopes have not been identified.

Population: Approximately 15 children with clinically diagnosed autism who have first degree relatives (parents, brothers, sisters, or children) with autoimmune disorders listed on a questionnaire. Children on the autism spectrum without autoimmune history and sibling matched controls without an ASD from the Simons Foundation Autism Research Initiative (SFARI) with deidentified data in the SFARI database will be matched for age, sex and ethnicity. Plasma samples and psychometric data from the database will be provided through the database for analysis in the laboratory of Dr. Reiter.

Design: The investigators seek to identify protein biomarkers in the serum of children with carefully characterized autism who have a familial autoimmune history in first degree relatives (FAH). Cognitive defects in the mouse model of the autism spectrum disorder tuberous sclerosis complex can be ameliorated by rapamycin, an immune suppressant drug indicating the likelihood that auto-immunity plays a role in autism pathogenesis. To expedite the identification of these biomarkers the investigators will use proteomic profiling in Drosophila melanogaster. The Drosophila (fly) nervous system is highly homologous to humans at the molecular level and genetic pathways for synaptic development and function are highly conserved. Several human neurogenetic diseases including Huntington, Alzheimer, fragile X, spinal cerebellar ataxia and Parkinson disease have been successfully studied using fly genetic models. Monoclonal antibodies generated against total fly brain homogenate cross react with human neuronal tissue and are highly specific for the recognition of particular subsets of neurons in the human nervous system. Our goal is to identify biomarkers in this group of autism patients, design a protein based assay system for screening serum for these biomarkers and confirm that these serum antibodies are persistent. A similar approach was taken by Dr. Levin to identify the central nervous system (CNS) autoantigen in the human T-lymphotropic virus type 1 disease associated myelopathy/tropical spastic. Dr. Reiter's group currently uses proteomic profiling in Drosophila to identify the protein targets of the Angelman syndrome gene, UBE3A.

ELIGIBILITY:
Inclusion Criteria:

* 4-17 years of age
* male or female
* autistic subjects must have a diagnosis of autism spectrum disorder

Exclusion Criteria:

* Controls must have no diagnosis of autism spectrum disorder.
* controls must be typically developing children without behavioral deviations.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with or without autism
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-11; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of autistic participants with autoimmune markers | 5 years
  The designed techniques will be used to first identify and then determine the frequency of autoimmune markers cross reacting with fly neuronal proteins in children with carefully characterized autism with and without a positive familial autoimmune history (FAH) in a first degree relative compared to typically developing children without FAH.

SECONDARY OUTCOMES:
Identification of neuronal protein autoimmunity | 5 years
  Presence of autoantibodies will be correlated with presence of a positive FAH in a first degree relative. Identification of neuronal protein autoimmunity will allow further investigation of etiological factors and possible immune modulating treatment in children with autism.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A McVicar, MD, Principal Investigator — LeBonheur Children's Medical Center; Larry T Reiter, PhD, Principal Investigator — LeBonheur Children's Medical Center
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided